CLINICAL TRIAL: NCT04373408
Title: Does Anterolateral Ligament Ultrasound Influences the Return-to-play After Anterior Cruciate Ligament Rupture? Survival Analysis
Brief Title: ALL Ultrasound Predicts the Success of ACL Repair?
Acronym: ALL_US
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Adrien Schwitzguebel (Other)
Responsible Party: Sponsor-Investigator, Adrien Schwitzguebel, MD, Hôpital de la Providence, Switzerland
Organization: Hôpital de la Providence, Switzerland (Other)
Other Study IDs: ALL Providence
Record Dates: First submitted 2020-04-30; First posted 2020-05-04 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Anterior Cruciate Ligament Rupture; Surgery
Keywords: Anterior Cruciate Ligament Rupture; Anterolateral ligament; Ultrasonography
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ACL rupture without indication for ALL surgery: Patients with an ACL rupture undergoing surgical repair of the ACL only
  Interventions: Procedure: ACL repair without anterolateral repair
- ACL rupture with indication for ALL surgery: Patients with an ACL rupture undergoing surgical repair of the ACL and the ALL
  Interventions: Procedure: ACL repair with anterolateral repair

INTERVENTIONS:
Procedure: ACL repair without anterolateral repair — Surgical repair of the ACL using semitendinous autograft
  Groups: ACL rupture without indication for ALL surgery
Procedure: ACL repair with anterolateral repair — Surgical repair of the ACL using semitendinous autograft, and surgical repair of the ALL using an allograft (Arthrex, Extra-Articular Augmentation device)
  Groups: ACL rupture with indication for ALL surgery

SUMMARY:
This case series evaluates whether patients with an anterior cruciate ligament (ACL) repair have better outcome if the anterolateral ligament (ALL) was repaired or not considering the ultrasound (US) pre-surgical recommendation.

DETAILED DESCRIPTION:
In this case series, the surgeon will decide which patient will have ACL only or ACL and ALL surgery on the basis on multiple parameters. All patient will undergo detailed pre-clinical evaluation, including an ultrasonographic evaluation of the integrity of the ALL.

Two subgroups will be compared for the primary outcome (International Knee Documentation Committee score at 8 months of follow-up). In subgroup 1, the surgeon will follow the ultrasonographic evaluation of the ALL considering the ALL repair (i.e. : ALL intact on the ultrasound, ACL repair only; ALL broken on ultrasound; ACL and ALL repair). In subgroup 2, the surgeon will not follow the ultrasonographic evaluation of the ALL considering the ALL repair.

Secondary outcomes of interest will be evaluated with multivariate regression analysis.

Sample size calculation:

The chosen parameter of interest for the primary outcome evaluation is a continuous response variable (IKDC score) from two independent subgroups (ultrasonographic evaluation of the ALL followed or not for the surgical repair), considering a ratio of 1:3 between the two subgroups. In a previous study (AJSM Sonnery-Cottet 2017) the response within each subject group was normally distributed with standard deviation 13.1. If the true difference between the group means is the published minimal clinically important difference of 9 (AJSM Nwachukwu 2017), we will need to study 30 experimental subjects and 90 control subjects to be able to reject the null hypothesis that the population means of the experimental and control groups are equal with probability (power) 0.9. The Type I error probability associated with this test of this null hypothesis is 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an ACL rupture and pre-surgical ultrasound evaluation

Exclusion Criteria:

* Sedentary patient without sports activities
* Prior ACL rupture of the same knee
* Posterior cruciate ligament rupture

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ACL rupture
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
IKDC score | Month 8
  Self-reported IKDC (International Knee Documentation Committee Subjective Knee Form) score, scaled between 0 and 100 (100 = good function)

SECONDARY OUTCOMES:
IKDC score | Months 0, 2, 5, 12
  Self-reported IKDC (International Knee Documentation Committee Subjective Knee Form) score, scaled between 0 and 100 (100 = good function)
Lysholm score | Months 0, 2, 5, 8, 12
  The Lysholm score is a 100-point scoring system for examining a patient's knee-specific symptoms including mechanical locking, instability, pain, swelling, stair climbing, and squatting, scaled between 0 and 100 (100 = good function)
SANE score | Months 0, 2, 5, 8, 12
  The Single Numeric Assessment Evaluation is a subjective percentage of the knee functionality, scaled between 0% and 100% (100% = good function)
Return-to-play | Months 5, 8, 12
  Timing when return-to-play to full sports activities is possible
Clinical evaluation: reverse pivot shift test | Months 0, 2, 5, 8, 12
  Described as "Clunk absent", "Clunk present", or "Clunk present with shake"
Clinical evaluation: anterior drawer test | Months 0, 2, 5, 8, 12
  Described as "Hard stop", "Soft stop", or "Soft stop and increased course"
Clinical evaluation: Lachman test | Months 0, 2, 5, 8, 12
  Described as "Hard stop", "Soft stop", or "Soft stop and increased course"
Clinical evaluation: thigh circumference 10 cm proximal to the patella | Months 0, 2, 5, 8, 12
  measure in cm
Clinical evaluation: thigh circumference 15 cm proximal to the patella | Months 0, 2, 5, 8, 12
  measure in cm
Clinical evaluation: knee extension | Months 0, 2, 5, 8, 12
  Measured in °. Negative values associated with bad outcome
Isokinetic test: knee extensors concentric strength | Months 5 & 8
  Measured in absolute value and comparative value with controlateral limb
Isokinetic test: knee flexors concentric strength | Months 5 & 8
  Measured in absolute value and comparative value with controlateral limb
Isokinetic test: knee flexors eccentric strength | Months 5 & 8
  Measured in absolute value and comparative value with controlateral limb
Rerupture rate | Year 3
  Patients will be evaluated by phone at 3 years of follow-up. Rerupture of the ACL graft (yes-no) will be recorded.

OTHER OUTCOMES:
Demographics: Age | Month 0
  Age of the patient (years)
Demographics: Sex | Month 0
  Sex of the patient
Demographics: timing between the trauma and the surgery | Month 0
  Time in days
Demographics: active tobacco use | Month 0
  binary outcome (yes - no)
Demographics: dyslipidemia | Month 0
  binary outcome (yes - no)
Demographics: past surgery of the knee | Month 0
  binary outcome (yes - no)
Demographics: Beighton score (joint hypermobility) | Month 0
  graded from 0 (no joint hypermobility) to 9 (major joint hypermobility)
Medial femorotibial chondropathy | Month 0
  Graded from 0 to 4 on arthroscopy
Lateral femorotibial chondropathy | Month 0
  Graded from 0 to 4 on arthroscopy
Femoropatellar chondropathy | Month 0
  Graded from 0 to 4 on arthroscopy
Internal lateral ligament tear | Month 0
  Described as "absent", "partial", or "full" on MRI
External lateral ligament tear | Month 0
  Described as "absent", "partial", or "full" on MRI
Internal meniscus lesion | Month 0
  Described as "absent", "present, not repaired", or "present, repaired" on arthroscopy
External meniscus lesion | Month 0
  Described as "absent", "present, not repaired", or "present, repaired" on arthroscopy
Surgical repair of the anterolateral ligament | Month 0
  Described as "not performed", or "performed" during surgery
Anterolateral ligament tear | Month 0
  Described as "intact", "partial tear", "full teat" or "non evaluable on ultrasonography

CONTACTS AND LOCATIONS:
Overall Officials: Adrien Schwitzguébel, MD, Principal Investigator — Hôpital de la Providence
Locations (1):
- Hôpital de la Providence, Neuchâtel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nwachukwu BU, Chang B, Voleti PB, Berkanish P, Cohn MR, Altchek DW, Allen AA, Williams RJ Rd. Preoperative Short Form Health Survey Score Is Predictive of Return to Play and Minimal Clinically Important Difference at a Minimum 2-Year Follow-up After Anterior Cruciate Ligament Reconstruction. Am J Sports Med. 2017 Oct;45(12):2784-2790. doi: 10.1177/0363546517714472. Epub 2017 Jul 20. PMID 28727937
- [Background] Sonnery-Cottet B, Saithna A, Cavalier M, Kajetanek C, Temponi EF, Daggett M, Helito CP, Thaunat M. Anterolateral Ligament Reconstruction Is Associated With Significantly Reduced ACL Graft Rupture Rates at a Minimum Follow-up of 2 Years: A Prospective Comparative Study of 502 Patients From the SANTI Study Group. Am J Sports Med. 2017 Jun;45(7):1547-1557. doi: 10.1177/0363546516686057. Epub 2017 Feb 2. PMID 28151693